CLINICAL TRIAL: NCT00743262
Title: Second Amendment on Phase I Trial NO7VEG 'Assessment of a Next Generation Indwelling Provox Voice Rehabilitation System (Vega)': Vega Siri Addendum.
Brief Title: Short-term Clinical Feasibility of the New Provox Vega 22.5 Voice Prosthesis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UD778
Record Dates: First submitted 2008-08-15; First posted 2008-08-28 (Estimated); Results first posted 2010-11-03 (Estimated); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Total Laryngectomy
Keywords: laryngectomy; larynx cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Provox voice prosthesis (Experimental)
  Interventions: Device: Provox voice prosthesis

INTERVENTIONS:
Device: Provox voice prosthesis — The current voice prosthesis (Provox ActiValve)of the patients will be removed and a new prosthesis (Provox Vega) will be inserted
  Other Names: Indwelling voice prosthesis

SUMMARY:
The purpose of this study is to investigate the performance of a new voice prosthesis in comparison with the Provox2 and the Provox ActiValve voice prosthesis in 15 laryngectomized patients. Factors taken into account are clinician and patient satisfaction with the insertion system, patient satisfaction with voice, speech, performance, and maintenance. Voice and speech will also be evaluated for the different prostheses by means of perceptual evaluations and acoustic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Total laryngectomy
* Use Provox ActiValve

Exclusion Criteria:

* Current problems with TE puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans JM Hilgers, MD, PhD, Principal Investigator — The Netherlands Cancer Institute; Michiel WM van den Brekel, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Provox Vega 22.5 French: A group of laryngectomized Provox ActiValve users tested the Provox Vega 22.5 French voice prosthesis for 3 weeks.
Period: Overall Study
Arm/Group | Provox Vega 22.5 French
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Provox Vega 22.5 French
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.33 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Region of Enrollment [Number; unit: patients]
  Netherlands | 15

OUTCOME MEASURES:

1. Primary Outcome: Short-term Feasibility Provox Vega 22.5 French
Description: Number of participants in whom the voice prosthesis was considered feasible in the short-term with regards to clinical and technical aspects as judged by patient and investigator.
Time Frame: 3 weeks
Measure: Number; unit: Patients
Arm/Group | Provox Vega 22.5 French
Number analyzed (Participants) | 15
Patients | 15

2. Secondary Outcome: Subjective Voice and Speech Quality
Description: Subjective participant opinion using a structured questionnaire addressing intelligibility face to face and on the phone, loudness, pitch and fluency. Each question was measured on a four point scale. Scores were summated, best possible score is 5, worst possible score is 20.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Provox Vega 22.5 French
Number analyzed (Participants) | 15
units on a scale | 6 (1.5)

3. Secondary Outcome: Device Life Time
Description: Device life time of the Provox Vega in days for replacement for leakage through the device. This is expected to be short (average about 3 weeks) since the Provox Vega 22.5 was tested in patients who normally use a Provox ActiValve. (Provox ActiValve is a problem solving prostheses used in patients who need frequent replacement of regular Provox voice prostheses short that are made of the same materials as the Provox Vega 22.5.)
Time Frame: one year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Provox Vega 22.5 French
Number analyzed (Participants) | 15
days | 39.7 (33)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the time the new Vega prosthesis was inserted until the voice prosthesis was replaced
Description: Adverse events were assessed after the insertion procedure, upon notification of a problem by the patient, and when the Provox Vega needed replacement. Normal reasons for replacement (leakage through, size changes) were not considered adverse events.
Arm/Group | Provox Vega 22.5 French
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Provox ActiValve users have short device life with normal indwelling prostheses (and hence use the Provox ActiValve). Therefore, the device life measured in this patient group is very short and not representative of the normal Provox Vega user.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No